CLINICAL TRIAL: NCT01338532
Title: Time to Total Hip Replacement in Patients With Hip Osteoarthritis Going Through Both Supervised Exercise and Patient Education Compared to Those Going Through Patient Education Only. A 3.5-6 Year Follow-up of a Randomized, Controlled, Clinical Trial.
Brief Title: Time to Total Hip Replacement After Supervised Exercise and Patient Education
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 03c-2011-NAR
Record Dates: First submitted 2011-04-18; First posted 2011-04-19 (Estimated); Last update posted 2012-08-20 (Estimated); Status verified 2012-08

CONDITIONS: Hip Osteoarthritis
Keywords: Hip osteoarthritis; Exercise; Patient Education; Total Hip Replacement
MeSH Terms: conditions — Osteoarthritis, Hip; Motor Activity | interventions — Patient Education as Topic

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Supervised exercise + patient education (Active Comparator)
  Interventions: Other: A 12 week supervised exercise program and patient education
- Patient education (Active Comparator)
  Interventions: Other: Patient education

INTERVENTIONS:
Other: A 12 week supervised exercise program and patient education — The exercise protocol included exercises from former studies on comparable patient populations. The intensity of the strength- and flexibility exercises meets the American College of Sports Medicine's (ACSM) recommendations for developing and maintaining muscular fitness in adults. Patients was required to exercise for approximately 60 minutes, to-three days a week for 12 weeks. Patient's attendance to the exercise program (compliance) was registered.
  All patients included in the study participated in a patient education program which included two individual and three small-group sessions lasting one hour each time.
  Arms: Supervised exercise + patient education
Other: Patient education — All patients included in the study participated in a patient education program which included two individual and three small-group sessions lasting one hour each time.
  Arms: Patient education

SUMMARY:
The purpose of this study is to evaluate the time to total hip replacement in patients with hip osteoarthritis going through both a supervised exercise program and patient education compared to patients going through patient education only.

The null hypothesis is: There are no differences in time to total hip replacement between patients with hip osteoarthritis who went through a 12 week supervised exercise program and patient education compared to patients who went through patient education only.

Material and methods:

109 patients with both symptomatically and radiographically verified hip osteoarthritis were included in this randomized controlled trial between april 2005 and october 2007. They were randomized to either a 12 week supervised exercise program and patient education (n=55) or patient education only (n=54).

Information on if and when total hip replacement is performed will be collected between April 1st and May 1st. Time since inclusion to follow-up will range from 3.5 to 6 years. Data will be collected directly from the study participants by telephone.

The main outcome is time to total hip replacement.

Status:

This study is a prolongation of an on-going RCT (3a-2005-NAR) using clinical outcomes to evaluate the effect of supervised exercise and patient education.

The study will be carried out: NAR-Department of Orthopedics, Ullevaal University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Between 40 and 80 years old with uni- or bilateral hip disability.
* Hip pain for more then 3 months.
* Harris Hip Score between 60 and 95. Harris Hip score (0-100 points) is widely used as an assessment of hip function in patients with hip OA. Harris Hip Score of 60 or below are used regularly at our institution as one of the criteria for total hip replacement surgery.
* Radiographic verified hip OA (Danielsson's criteria for radiographic OA: Danielsson's criteria for minimal joint space: < 4 mm < 70 years, < 3 mm ≥ 70 years, or 1 mm difference between hips).

Exclusion Criteria:

* Patients who have a history of resent trauma or functional impairment to the lower limbs or diseases which might interfere with participation (rheumatoid arthritis, cancer, osteoporosis, severe back pain, knee OA).
* Patients with co-morbidities not tolerating physical activities

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2005-03; Primary Completion 2013-05 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Time to Total Hip Replacement surgery (THR) | 3.5 to 6 years after inclusion
  All included patients will be examined regarding if they have gone through THR surgery since their inclusion in the present study. For those who report to have gone through THR surgery, date for when surgery were performed will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: May Arna Risberg, PT, PhD, Principal Investigator — NAR- Department of Orthopedics, Oslo University Hospital
Locations (1):
- NAR-Orthopedic Department, Oslo University Hospital & Hjelp24 NIMI, Oslo, Norway

REFERENCES:
- [Derived] Svege I, Nordsletten L, Fernandes L, Risberg MA. Exercise therapy may postpone total hip replacement surgery in patients with hip osteoarthritis: a long-term follow-up of a randomised trial. Ann Rheum Dis. 2015 Jan;74(1):164-9. doi: 10.1136/annrheumdis-2013-203628. Epub 2013 Nov 19. PMID 24255546
- See also: Homepage NAR — http://www.active-rehab.no